CLINICAL TRIAL: NCT01410279
Title: Inspiratory Muscle Training Effect on the Functional Capacity and the Quality of Life in Chronic Pulmonary Hypertension
Brief Title: Inspiratory Muscle Training in Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Pedro Dal'Lago, UFCSPA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09032
Record Dates: First submitted 2011-04-20; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; inspiratory muscle training; inspiratory muscle weakness; pulmonary functional; functional capacity; quality of life
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Inspiratory muscle training — The load is adjusted weekly in thirty percent of maximal inspiratory pressure of the subject.

SUMMARY:
The purpose of this study is evaluate the effect the inspiratory muscle training on the functional capacity of patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a syndrome, in the case of hemodynamic alteration of a number of diseases and processes, such as the progressive increase in pulmonary vascular resistance, right heart failure and early death. Frequently patients with PH have reduced functional capacity, quality of life and survival. It was demonstrated recently that patients with HP also have inspiratory muscle weakness, possibly further increase the fatigue and dyspnea during exercise. To meet this need, inspiratory muscle training can lead to significant improvement in respiratory muscle strength, exercise tolerance and dyspnea, thus resulting in reduction of discomfort during activities of daily living, increase in exercise capacity and improved quality of life in different situations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis pulmonary hypertension
* World Health Organization (WHO) functional class II to IV
* inspiratory muscle weakness

Exclusion Criteria:

* obesity
* chronic obstructive pulmonary disease
* orthopedic and neurological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The distance traveled in meters in the six minutes walk test after 8 weeks the inspiratory muscle training | patients will be monitored throughout the training protocol for 8 weeks

SECONDARY OUTCOMES:
Increase in score of quality of life questionnaire after 8 weeks the inspiratory muscle training | patients will be monitored throughout the training protocol for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Dal'Lago, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinica de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941